CLINICAL TRIAL: NCT02923856
Title: A Multi-center Study for Eradication of Helicobacter Pylori With Triple Therapy Based on Accurate Susceptibility Testing of Clarithromycin
Brief Title: A Multi-center Study for Eradication of Helicobacter Pylori With Triple Therapy Using Clarithromycin
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sanmen People's Hospital (Other)
Collaborators: Wenzhou Central Hospital (Other); The First Affiliated Hospital with Nanjing Medical University (Other); Taizhou Hospital (Other); Affiliated Wenling Hospital of Wenzhou Medical University (Other); Hangzhou Medical College (Other); Centers for Disease Control and Prevention, China (Other Government); Zhiyuan Medical Inspection Institute (Other)
Responsible Party: Principal Investigator, Hongzhang Li, Director of Sanmen People's Hospital, Sanmen People's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SanmenPH
Record Dates: First submitted 2016-08-23; First posted 2016-10-05 (Estimated); Last update posted 2019-02-19 (Actual); Status verified 2018-08

CONDITIONS: Gastritis
Keywords: Helicobacter pylori; Antibiotic resistance; Sequencing
MeSH Terms: conditions — Gastritis

ARMS (7):
- Clarithromycin resistance group (Experimental): Patients who are resistant to clarithromycin in susceptibility test were classified into clarithromycin resistance group.
  Interventions: Device: The results of clarithromycin susceptibility test of H. pylori isolates
- 7 days Successful treatment (Experimental): The successful treatment of H. pylori group were treatment successful patients after the 7days standardized treatment.
  Interventions: Device: The results of clarithromycin susceptibility test of H. pylori isolates; Device: Computer generated random number, randomly assigned into groups; Device: The result of 13C-urea breath test of patient in 7days/10days/14days treatment groups
- 7 days failed treatment (Experimental): The failed treatment of H. pylori group were treatment failure patients after the 7days standardized treatment.
  Interventions: Device: The results of clarithromycin susceptibility test of H. pylori isolates; Device: Computer generated random number, randomly assigned into groups; Device: The result of 13C-urea breath test of patient in 7days/10days/14days treatment groups
- 10 days Successful treatment (Experimental): The successful treatment of H. pylori group were treatment successful patients after the 10days standardized treatment.
  Interventions: Device: The results of clarithromycin susceptibility test of H. pylori isolates; Device: Computer generated random number, randomly assigned into groups; Device: The result of 13C-urea breath test of patient in 7days/10days/14days treatment groups
- 10 days failed treatment (Experimental): The failed treatment of H. pylori group were treatment failure patients after the 10days standardized treatment.
  Interventions: Device: The results of clarithromycin susceptibility test of H. pylori isolates; Device: Computer generated random number, randomly assigned into groups; Device: The result of 13C-urea breath test of patient in 7days/10days/14days treatment groups
- 14 days Successful treatment (Experimental): The successful treatment of H. pylori group were treatment successful patients after the 14days standardized treatment.
  Interventions: Device: The results of clarithromycin susceptibility test of H. pylori isolates; Device: Computer generated random number, randomly assigned into groups; Device: The result of 13C-urea breath test of patient in 7days/10days/14days treatment groups
- 14 days failed treatment (Experimental): The failed treatment of H. pylori group were treatment failure patients after the 14days standardized treatment.
  Interventions: Device: The results of clarithromycin susceptibility test of H. pylori isolates; Device: Computer generated random number, randomly assigned into groups; Device: The result of 13C-urea breath test of patient in 7days/10days/14days treatment groups

INTERVENTIONS:
Device: The results of clarithromycin susceptibility test of H. pylori isolates — According to the results of antibiotic susceptible testing, patients who were resistant to clarithromycin were belonged into clarithromycin resistance group.Patients who were sensitive to clarithromycin were belonged into the 7days/10days/14days treatment groups.
Device: Computer generated random number, randomly assigned into groups — The patients with clarithromycin sensitive. Computer generated random number,randomly assigned into 7days/10days/14days treatment groups.
  Arms: 10 days Successful treatment; 10 days failed treatment; 14 days Successful treatment; 14 days failed treatment; 7 days Successful treatment; 7 days failed treatment
Device: The result of 13C-urea breath test of patient in 7days/10days/14days treatment groups — The intervention focused on the results from the result of 13C-urea breath test at 8 weeks after treatment in patients. All patients were taking 75mg 13C-urea and analysis with a modified isotope ratio mass spectrometer to determine the 13CO2 content.The successful treatment groups were patients with negative in 13C-urea breath tests.The failed treatment of H. pylori groups were patients with positive in 13C-urea breath tests after the standardized triple therapy treatment.
  Arms: 10 days Successful treatment; 10 days failed treatment; 14 days Successful treatment; 14 days failed treatment; 7 days Successful treatment; 7 days failed treatment

SUMMARY:
As the resistant rate of the Helicobacter pylori to some common antibiotics was rising，the eradication rate of the Helicobacter pylori with the standard triple therapy failed to exceed 70% in China，and had to drop out of the first-line treatment recommendations. However, with the increase of treatment time, patients burden, adverse reactions of antibiotics or proton pump inhibitor (PPI) will also increase. Resistance to clarithromycin is the major cause of the failure to eradicate Helicobacter pylori. But, in terms of population, there are still more than 70% of the patients with clarithromycin sensitive. Under the guidance with susceptibility test，7-day standard triple therapy could be used. In this study, investigators will select the patients with infection of H. pylori and with clarithromycin sensitive. Eradication of Helicobacter pylori with triple therapy based on accurate susceptibility testing of clarithromycin will be studied. The treatment time will be assigned into 7 days,10 days and 14 days groups. Then, investigators will perform a sequencing for failed treatment patients in groups, such as drug resistance gene mutation, phenotype and genotype. Finally, investigators will compare the differences between the patients with triple therapy and traditional quadruple therapy.The incidence of adverse effects in the eradicate treatment will reduce at least 10% and avoid patients' unnecessary economic losses at least 400RMB per person.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18~70 years old, male or female, the first eradication therapy of H. pylori infection patients.
2. Symptoms of abdominal pain, bloating, acid efflux, belching, nausea, vomiting, heartburn, chest pain, vomiting, melena, etc.
3. Unused antibiotics, bismuth, H2 receptor antagonists or PPI by nearly 4 weeks
4. 13C-labelled urea breath test positive.
5. Agreed to Helicobacter pylori culture and sensitivity testing taken by endoscopy gastric biopsy specimens,and the result of culture was positive.
6. Agreed to Helicobacter pylori eradication therapy and cooperate with the eradication efficacy follow-up survey.

Exclusion Criteria:

1. Severe heart, liver, kidney dysfunction.
2. Pregnant or lactating women.
3. Complications of bleeding, perforation, pyloric obstruction, cancer.
4. Within 3 months before with the drugs involved in other drugs research.
5. Esophageal,gastrointestinal surgery history.
6. Patients can not properly express their complaints,such as psychosis, severe neurosis.
7. Taking NSIAD or alcohol abusers.
8. Allergic to amoxicillin or clarithromycin tested by susceptibility testing.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 672 (Estimated)
Dates: Start 2017-01; Primary Completion 2019-12 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
The accurate determination of clarithromycin susceptibility. | 2 years
  Assess bacterial susceptibility to antibiotics using the agar diffusion method. The Resistance point of clarithromycin was divided into 0.125μg/ml,0.25μg/ml,0.5μg/ml and 1μg/ml.Test clarithromycin resistance of Helicobacter pylori for patients.
Establish individualized precision triple therapy based on minimal inhibitory concentration. | 2.5 years
  Based on the clarithromycin accurate susceptibility，pinpoint different courses of triple treatment therapy targeted to different people based on minimal inhibitory concentration of clarithromycin.

SECONDARY OUTCOMES:
The incidence of adverse effects | 3 years
  Drugs targeted, it could reduce the intake of antibiotics for patients.The incidence of adverse effects in the eradicate treatment will reduce. Avoid patients' unnecessary economic losses.

OTHER OUTCOMES:
Impact of mixed infection and CYP2C19 genotype on eradication rate for Helicobacter pylori with triple therapy using clarithromycin. | 3 years
  Investigators will perform a sequencing for failed treatment patients in groups, such as drug resistance gene mutation,and CYP2C19 genotype. Evaluating the impact of mixed infection and CYP2C19 genotype on eradication rate for Helicobacter pylori with triple therapy.

CONTACTS AND LOCATIONS:
Locations (1):
- Sanmen People's hospital, Taizhou, Zhejiang, China